CLINICAL TRIAL: NCT05791552
Title: Feasibility of a Method for Analysis of Alzheimer´s Disease Specific Proteins in Nasal Secretion
Acronym: NL02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Noselab GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MUC-00
Record Dates: First submitted 2023-03-14; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Nasal Secretion; Alzheimer Disease; Brain Nose Interface
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Patient WITH cognitive impairment and no nasal pathologies. CSF analysis is planned or results are already available
  Interventions: Diagnostic Test: Collection of nasal secretion
- Group B (Other): Patient WITHOUT cognitive impairment and without nasal pathologies
  Interventions: Diagnostic Test: Collection of nasal secretion

INTERVENTIONS:
Diagnostic Test: Collection of nasal secretion — Standardized collection of nasal secretion in the vicinity of the olfactory cleft

SUMMARY:
This study is a first in man study investigating the feasibility of the collection, storage, processing and analysis of 4 key biomarkers for the diagnosis of Alzheimer's disease [AD] in nasal secretion. Nasal secretion [NS] constitutes a minimally invasive access to cerebrospinal fluid [CSF]. Therefore, it could be highly suitable for detection and monitoring of the AD relevant biomarkers pTau181, total Tau, Amyloid-ß1-40 and Amyloid-ß1-42. This study evaluates correlations of biomarker patterns in NS and CSF. Furthermore, the correlations of the 4 AD specific biomarkers in nasal secretion and CSF is investigated. For this study, patients with cognitive impairment (AD and NonAD group) and healthy controls were included.

ELIGIBILITY:
Inclusion Criteria:

* Group A Patient WITH cognitive impairment and no nasal pathologies. CSF analysis is planned or results are already available
* Group B Patient WITHOUT cognitive disorder and without pathologies in the nasal area

Exclusion Criteria:

* Presence of an obstructing nasal cavity disease
* Patient suffers from an acute upper respiratory tract infection (putrid rhinorrhea)
* Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Detection of brain specific biomarkers in nasal secretion | 1-2 years
  The aim of the study was to investigate the overall applicability of a new, minimally invasive, and proprietary procedure developed by the company Noselab GmbH for exclusion or detection of Alzheimer's disease (AD) and/or neurodegeneration (ND) in patients with (subjective) cognitive impairment.
Distinction of pathologic and physiologic biomarker patterns in nasal secretion | 1-2 years
  Assess ranges of biomarkers for AD in nasal secretion of cognitively impaired patients with and without AD and healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- Noselab GmbH, München, Bavaria, Germany